CLINICAL TRIAL: NCT00829218
Title: A Clinical Trial Examining the Effects of the Food Additive Glutamate on Irritable Bowel Syndrome and Fibromyalgia
Brief Title: Clinical Trial Examining Effects of Monosodium Glutamate (MSG) on Irritable Bowel Syndrome (IBS) and Fibromyalgia (FM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Principal Investigator, Kathleen F. Holton, Research Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 4763
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Irritable Bowel Syndrome; Fibromyalgia
Keywords: Irritable Bowel Syndrome; Fibromyalgia; Glutamate; Diet; Food additives
MeSH Terms: conditions — Irritable Bowel Syndrome; Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Glutamate challenge (Active Comparator): Glutamate challenge: After the one month glutamate free diet, subjects will receive 5 grams of glutamate for three days on one week and placebo for three days on the next week. Arm 1 is the 5 grams of glutamate which will be given in a mixed juice.
  Interventions: Other: Glutamate additive-free diet
- 2- Placebo (Placebo Comparator): Glutamate challenge: After the one month glutamate free diet, subjects will receive 5 grams of glutamate for three days on one week and placebo for three days on the next week. Arm 2 is the placebo arm, which will be juice with nothing added.
  Interventions: Other: Glutamate additive-free diet; Other: Placebo diet

INTERVENTIONS:
Other: Glutamate additive-free diet — All subjects will follow a diet for one month where all foods containing the additive glutamate have been removed. At the end of the one month diet, subjects who have responded positively to the diet will go onto the challenge arms of the study, where they will be randomized to receive placebo (mixed juice alone) for three days on one week, and 5 grams of glutamate in the mixed juice for three days on the other week.
  Other Names: Glutamate will be used as a challenge in the form of MSG.
Other: Placebo diet — Juice with nothing added.
  Arms: 2- Placebo

SUMMARY:
Objective: Randomized, double blind, placebo-controlled, crossover, clinical trial to examine the effects of the food additive glutamate (in the form of MSG) on IBS and fibromyalgia.

Setting and Subjects: The Fibromyalgia Research Database at OHSU will be utilized to identify and recruit fibromyalgia patients who also have IBS to OHSU study centers.

Intervention: Approximately 60 male and female subjects aged 18-75 will be placed on a 1-month glutamate-free elimination diet. Those that respond positively to the diet (we are estimating 30-40 subjects), will then be randomized to receive either a citrus drink containing 5 grams of MSG; or placebo (the citrus drink alone)on three consecutive days one week apart.

The investigators are hypothesizing that those who react positively to the elimination diet will have symptom occurrence statistically more frequently when given the glutamate challenge, than when given placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-75 who fulfill criteria for Irritable Bowel Syndrome (IBS) and Fibromyalgia (FM)
* They must live in the greater Portland, OR, metro area, have transportation to/from study site, have access to email
* Willing to discontinue medications with bowel altering side effects

Exclusion Criteria:

* Asthma
* Inflammatory bowel disease
* Colon cancer or active endometriosis
* Any major abdominal surgery (excluding caesarean section, tubal ligation, hernia repair, gall bladder removal or appendectomy)
* Female and pregnant
* Currently taking pregabalin, gabapentin, or anti-psychotic medications and are unwilling/ unable to discontinue use
* Suffered from alcohol/substance abuse or psychosis in the last two years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the number of patients who have a positive response to a one month glutamate free diet, as measured by the Perception of Global Impression of Change (PGIC) scores | 4 weeks
To assess whether symptoms return with MSG challenge statistically more frequently than with placebo as measured by symptom scores. | 6 weeks, 7 weeks

SECONDARY OUTCOMES:
Improvement on Irritable Bowel Syndrome-Quality of Life (IBS-QOL) questionnaire | 4 weeks, 7 weeks
Improvement in day-to-day functioning based on the Revised Fibromyalgia Impact Questionnaire | 4 weeks, 7 weeks
A reduction in pain based on two visual analog scales, one for gut pain, and another for musculo-skeletal pain | 4 weeks, 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Taren, PhD, Study Chair — University of Arizona; Kathleen F Holton, MPH, PhDc, Principal Investigator — University of Arizona and Oregon Health & Science Univ.; Kimberly D Jones, PhD, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Holton KF, Taren DL, Thomson CA, Bennett RM, Jones KD. The effect of dietary glutamate on fibromyalgia and irritable bowel symptoms. Clin Exp Rheumatol. 2012 Nov-Dec;30(6 Suppl 74):10-7. Epub 2012 Dec 14. PMID 22766026